CLINICAL TRIAL: NCT00107250
Title: A Phase I, Open-Label, Dose-Seeking Study of AZD2171 Given Daily Orally in Combination With Standard Chemotherapy Regimens (CT) in Patients With Advanced Incurable Non-Small Cell Lung Cancer (NSCLC) or Colorectal Cancer or Other Tumor Types Suitable for Treatment With Capecitabine
Brief Title: AZD2171 + Chemotherapy in Advanced NSCLC, Colorectal Cancer, or Other Cancer Suitable for Treatment With Capecitabine (Non-Small Lung Cancer Patients Closed to Enrollment as 8/9/07)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I171; CAN-NCIC-IND171 (Other: PDQ); CDR0000422357 (Other: PDQ)
Record Dates: First submitted 2005-04-05; First posted 2005-04-06 (Estimated); Last update posted 2023-08-04 (Actual); Status verified 2020-04

CONDITIONS: Colorectal Cancer; Lung Cancer; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: recurrent non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; stage IV colon cancer; stage IV rectal cancer; unspecified adult solid tumor, protocol specific
MeSH Terms: conditions — Colorectal Neoplasms; Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Colonic Neoplasms; Rectal Neoplasms | interventions — Capecitabine; Carboplatin; cediranib; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AZD2171 + Standard chemotherpay regimens (Experimental)
  Interventions: Drug: capecitabine; Drug: carboplatin; Drug: cediranib maleate; Drug: paclitaxel

INTERVENTIONS:
Drug: capecitabine — 1000 mg/m2 orally twice daily (total of 2000 mg/m2 per day) for the first 14 days of a 21 day cycle for a maximum of 6-8 cycles.
Drug: carboplatin — AUC 6; IV; 30 minutes; Every 21 days for a maximum of 6-8 cycles
Drug: cediranib maleate — Given daily; orally with approximately 240 ml of water whilst in an upright position
Drug: paclitaxel — 200mg/m2; IV; 3 hours; Every 21 days for a maximum of 6-8 cycles

SUMMARY:
RATIONALE: AZD2171 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Drugs used in chemotherapy, such as paclitaxel, carboplatin, or capecitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving AZD2171 together with chemotherapy may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of AZD2171 when given together with chemotherapy in treating patients with advanced non-small cell lung cancer (closed to enrollment as of 8/9/07), colorectal cancer, or other cancer suitable to capecitabine treatment.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose and recommended phase II dose of AZD2171 when administered in combination with standard chemotherapy comprising either paclitaxel and carboplatin OR capecitabine in patients with advanced incurable non-small cell lung cancer (closed to accrual as of 8/9/07), colorectal cancer, or other tumor types suitable for treatment with capecitabine.
* Determine the safety and tolerability of these regimens in these patients.
* Determine the toxicity profile and dose-limiting toxic effects of these regimens in these patients.
* Determine the pharmacokinetic profile of these regimens in these patients.
* Correlate the toxicity profile with the pharmacokinetic profile of these regimens in these patients.
* Determine the antitumor activity of these regimens in patients with measurable disease.
* Correlate patient outcome (response) with baseline (using tumor samples) and serial (using urine and plasma samples) biomarkers in patients treated with these regimens.

OUTLINE: This is an open-label, multicenter, dose-escalation study of AZD2171. Patients are assigned to 1 of 2 treatment groups according to diagnosis.

* Group 1 (non-small cell lung cancer) (closed to accrual as of 8/9/07): Patients receive paclitaxel IV and carboplatin IV on day 1. Patients also receive oral AZD2171 once daily on days 2-21 of course 1 and on days 1-21 of all subsequent courses. Treatment with paclitaxel and carboplatin repeats every 21 days for up to 8 courses in the absence of disease progression or unacceptable toxicity. Treatment with AZD2171 repeats every 21 days in the absence of disease progression or unacceptable toxicity.
* Group 2 (colorectal or other tumor types): Patients receive oral capecitabine twice daily on days 1-14. Patients also receive oral AZD2171 once daily on days 8-21 of course 1 and on days 1-21 of all subsequent courses. Treatment with capecitabine repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Treatment with AZD2171 repeats every 21 days in the absence of disease progression or unacceptable toxicity.

In both groups, patients achieving a complete response (CR) OR a stable partial response (SPR) receive 2 additional courses beyond CR or SPR.

Cohorts of 3-6 patients per group receive escalating doses of AZD2171 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity. Up to 30 additional patients (20 in group 1 and 10 in group 2) will be treated at the MTD.

After completion of study treatment, patients are followed at 4 weeks and then every 3 months until disease relapse.

PROJECTED ACCRUAL: A total of 3-35 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed diagnosis of 1 of the following:

  * Non-small cell lung cancer (NSCLC) (closed to accrual as of 8/9/07) meeting 1 of the following stage criteria:

    * Stage IIIB disease

      * Patients without pleural effusion who are not candidates for combined modality treatment OR who were treated at centers where combined modality treatment is not considered standard treatment are eligible
    * Stage IV disease
    * Local or metastatic failure after prior surgery and/or radiotherapy
  * Colorectal cancer

    * Metastatic disease
    * Considered suitable for first-line therapy with capecitabine
  * Other tumor types

    * Suitable for treatment with capecitabine
    * No more than 2 prior chemotherapy regimens for advanced or metastatic disease
* Incurable by radiotherapy or surgery
* Clinically or radiologically documented disease

  * No tumor marker elevation as the only evidence of disease
* No necrotic or hemorrhagic tumor or metastases
* No untreated brain or meningeal metastases

  * Patients with previously treated stable brain metastases (by radiography or clinical exam) are eligible provided they are asymptomatic and do not require corticosteroids

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* At least 12 weeks (colorectal cancer patients)

Hematopoietic

* Hemoglobin adequate

  * Anemia allowed provided patient is well compensated with no evidence of recent bleeding
* Absolute granulocyte count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* No overt bleeding (i.e., ≥ 30 mL/episode) within the past 3 months

Hepatic

* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* ALT or AST ≤ 2 times ULN (5 times ULN for documented liver metastases)

Renal

* Creatinine ≤ 1.5 times ULN OR
* Creatinine clearance ≥ 50 mL/min
* No proteinuria > grade 1

Cardiovascular

* Resting systolic blood pressure ≤ 150 mm Hg AND/OR resting diastolic blood pressure ≤ 100 mm Hg (in the presence or absence of a stable dose of antihypertensive medication)
* Mean QTc ≤ 470 msec (with Bazetts correction) by ECG
* LVEF > 50% for patients with prior anthracyclines/trastuzumab or cardio-toxic agents
* No untreated or uncontrolled cardiovascular condition
* No symptomatic cardiac dysfunction
* No poorly controlled hypertension
* No history of labile hypertension
* No history of poor compliance with antihypertensive medication
* No history of familial long QT syndrome

Pulmonary

* No clinically relevant hemoptysis (i.e., ≥ 5 mL fresh blood) within the past 4 weeks

  * Patients with only flecks of blood in their sputum are eligible

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective (double-method for females; barrier method for males) contraception
* No prior allergic reaction to drugs containing Cremophor EL® (NSCLC patients [closed to accrual as of 8/9/07])
* No peripheral neuropathy > grade 1 (NSCLC patients [closed to accrual as of 8/9/07])
* No dihydropyrimidine dehydrogenase deficiency (colorectal cancer patients)
* No history of severe hand-foot syndrome after treatment with fluoropyrimidines (colorectal cancer patients)
* No other malignancy within the past 5 years except adequately treated nonmelanoma skin cancer or other curatively treated solid tumor
* No active or uncontrolled infection
* No other serious illness or medical condition that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior antiangiogenesis therapy

Chemotherapy

* At least 4 weeks since prior single-agent non-platinum-containing chemotherapy (6 weeks for nitrosoureas or mitomycin) for metastatic disease (NSCLC patients [closed to accrual as of 8/9/07])

  * No more than 1 prior single-agent non-platinum-containing chemotherapy regimen for metastatic disease
* At least 6 months since prior adjuvant or neoadjuvant chemotherapy
* No prior taxane therapy (NSCLC patients [closed to accrual as of 8/9/07])
* No prior chemotherapy for metastatic disease (colorectal cancer patients)
* No prior capecitabine (colorectal cancer patients)

Endocrine therapy

* See Disease Characteristics
* At least 4 weeks since prior corticosteroids

Radiotherapy

* See Disease Characteristics
* At least 21 days since prior palliative radiotherapy except for low-dose non-myelosuppressive radiotherapy with approval
* At least 6 months since prior adjuvant radiotherapy

Surgery

* See Disease Characteristics
* At least 14 days since prior major surgery

Other

* Recovered from prior therapy
* At least 14 days since prior epidermal growth factor receptor inhibitor therapy
* Concurrent oral anticoagulants (e.g., warfarin) allowed provided INR is strictly monitored
* No other concurrent investigational therapy
* No other concurrent anticancer therapy
* No concurrent prophylactic pyridoxine (vitamin B_6) for hand-foot syndrome (colorectal or other tumor type patients)

  * Use of pyridoxine after the onset of hand-foot syndrome allowed at the discretion of the physician

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2005-01-21 (Actual); Primary Completion 2009-10-23 (Actual); Study Completion 2011-01-18 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity | Each dose level
  To recommend phase II dose of AZD2171 when given orally daily in combination with standard chemotherapy in patients with advanced NSCLC or colon cancer or other tumour types suitable for treatment with capecitabine.

SECONDARY OUTCOMES:
Safety | Each dose level
  safety, tolerability, toxicity profile, dose limiting toxicities and pharmacokinetic profile of AZD2171 and standard chemotherapy given in these combinations. The correlation, if any,between the toxicity profile and the pharmacokinetics will be determined.
Anti-tumour activity | Each dose level
  Assessing the anti-tumour activity of AZD2171 in combination with standard chemotherapy regimens in patients with measurable disease.
Tumour Response | Each dose level
  To correlate patient outcomes (response) with baseline (tumour) and serial (urine and plasma) biomarkers

CONTACTS AND LOCATIONS:
Overall Officials: Derek Jonker, MD, Study Chair — Ottawa Regional Cancer Centre; Scott A. Laurie, MD, FRCPC, Study Chair — Ottawa Regional Cancer Centre
Locations (2):
- Canada (2):
  - Ottawa Hospital Regional Cancer Centre - General Campus, Ottawa, Ontario
  - Princess Margaret Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Laurie SA, Gauthier I, Arnold A, Shepherd FA, Ellis PM, Chen E, Goss G, Powers J, Walsh W, Tu D, Robertson J, Puchalski TA, Seymour L. Phase I and pharmacokinetic study of daily oral AZD2171, an inhibitor of vascular endothelial growth factor tyrosine kinases, in combination with carboplatin and paclitaxel in patients with advanced non-small-cell lung cancer: the National Cancer Institute of Canada clinical trials group. J Clin Oncol. 2008 Apr 10;26(11):1871-8. doi: 10.1200/JCO.2007.14.4741. PMID 18398152